CLINICAL TRIAL: NCT02141893
Title: Effectiveness of a Multi-level Clinic and Family Asthma Intervention With a Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Glorisa Canino, Glorisa Canino, University of Puerto Rico
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GC- 0160609-CALMA; P60MD00226 (Other Grant/Funding Number: National Center on Minority Health and Health Disparities)
Record Dates: First submitted 2014-05-12; First posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Infantile Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CALMA (Active Comparator): Participants only received a family education intervention (previously tested) known as CALMA
  Interventions: Behavioral: CALMA plus; Behavioral: CALMA
- Calma plus (Experimental): Participants in Arm 2 received the CALMA family education intervention and physician education and organizational change of the clinics were addressed with a culturally tailored program developed by adapting content from several evidence-based provider training programs.
  Interventions: Behavioral: CALMA plus

INTERVENTIONS:
Behavioral: CALMA plus — Participants received a family education intervention (previously tested) known as CALMA plus physician education and organizational change of the clinics were addressed with a culturally tailored program developed by adapting content from several evidence-based provider training programs
Behavioral: CALMA — Family Education Intervention on management of pediatric asthma
  Arms: CALMA

SUMMARY:
The aim of this group-randomized trial was to test the effectiveness of a new comprehensive program, which the investigators called CALMA -plus, in increasing controller medication use and reducing asthma symptoms. CALMA-plus involved the CALMA home-based family intervention, plus educational training of physicians and nurses, as well as screening for asthma in clinics serving Medicaid island Puerto Rican children with asthma. Because the provider training was expected to have an impact on the entire clinical setting where trained providers work, as well as the patients using that setting, the investigators randomized clinic groups rather than individual patients. The investigators compared the CALMA-Plus intervention to a CALMA-only group, which the investigators expected to obtain the same benefits as the investigators have previously documented.

DETAILED DESCRIPTION:
Puerto Rico has high rates of pediatric asthma and morbidity associated in part with poor family asthma management and low rates of controller medication use. A previous study found a family management intervention called CALMA to be effective in reducing asthma symptoms and service utilization. However, CALMA was not effective in increasing the use of controller medications. CALMA- plus was developed to address this issue by adding to CALMA components of educational training of physicians and nurses, and screening for asthma in clinics serving Medicaid Puerto Rican children with persistent asthma. A total of 404 children in eight clinics were studied after forming four pairs of clinics and randomizing the clinics (1:1) to CALMA-only or CALMA-plus within each pair. After adjusting for clinic variation, the study failed to demonstrate that the CALMA-plus intervention was more efficacious than the CALMA- only intervention for increasing reported controller medication use or decreasing symptoms in children with persistent asthma. Both groups had lower rates of asthma symptoms and service utilization consistent with previous results of the CALMA-only intervention. Limitations of the study were small number of clinics available, comparison of the experimental intervention with an evidence based intervention, and limited exposure to some aspects of the intervention. More effective interventions may include aggressive case management, and providing the physician with more relevant information.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria required that the child have at least one claim with a diagnostic code for asthma or reactive airway disease (International Classification of Diseases (ICD 9) diagnostic code 493.xx) and in the last year period had either1) been hospitalized for asthma
* had at least 2 Emergency Department (ED) visits
* 3-5 ambulatory visits due to asthma
* utilized asthma medications from 2 of the following therapeutic categories: Anticholinergics, cromolyn, sympathomimetics, steroid inhalants, methylxanthines, leukotriene inhibitors, or corticosteroids.

Exclusion Criteria:

* currently participating in another asthma study
* no appropriate address for follow-up in the claims data.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 404 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in Percentage of participants using controller medications for asthma from baseline to 12 month follow-up | Baseline, 12

SECONDARY OUTCOMES:
Change in the Reduction of asthma symptomatology from baseline to 12 month follow-up | baseline, 12

CONTACTS AND LOCATIONS:
Overall Officials: Glorisa Canino, PhD, Principal Investigator — Medical Sciences Campus
Locations (1):
- Behavioral Sciences Research Institute, San Juan, PR, Puerto Rico

REFERENCES:
- [Derived] Canino G, Shrout PE, Vila D, Ramirez R, Rand C. Effectiveness of a multi-level asthma intervention in increasing controller medication use: a randomized control trial. J Asthma. 2016;53(3):301-10. doi: 10.3109/02770903.2015.1057846. Epub 2016 Jan 19. PMID 26786240